CLINICAL TRIAL: NCT03660930
Title: A Phase 1/2 Study of Nab-Sirolimus With Pazopanib (VOTRIENT®) in Patients With Advanced Nonadipocytic Soft-Tissue Sarcomas
Brief Title: Nab-Sirolimus and Pazopanib Hydrochloride in Treating Patients With Advanced Nonadipocytic Soft Tissue Sarcomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated at completion of the Phase 1 dose escalation due to loss of financial support.
Sponsor: University of Washington (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Principal Investigator, Lee Duncan Cranmer, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1718053; 10015 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2018-01624 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced Soft Tissue Sarcoma; Locally Advanced Soft Tissue Sarcoma; Metastatic Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ABI-009, pazopanib) (Experimental): Participants receive nab-sirolimus intravenously (IV) on days 1 and 8 or day 1 only and pazopanib hydrochloride orally (PO) daily on days 1-21. Cycles repeat every 21 days until unequivocal clinical disease progression, unacceptable toxicity, or until in the opinion of the investigator the patient is no longer benefiting from therapy, or at the patient's discretion.
  Interventions: Drug: Sirolimus Albumin-bound Nanoparticles; Drug: Pazopanib hydrochloride

INTERVENTIONS:
Drug: Sirolimus Albumin-bound Nanoparticles — Given IV
  Other Names: Nab-Rapamycin; Nanoparticle Albumin-Bound Rapamycin; ABI-009; Nanoparticle Albumin-bound Sirolimus; Fyarro; Sirolimus Protein-bound Particles
Drug: Pazopanib hydrochloride — Given PO
  Other Names: Votrient

SUMMARY:
This phase I/II trial studies the side effects and best dose of nab-sirolimus and how well it works when given together with pazopanib hydrochloride in treating participants with nonadipocytic soft tissue sarcomas that has spread to other places in the body (advanced). Nab-sirolimus and pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of nanoparticle albumin-bound rapamycin followed by a phase II study.

Participants receive nab-sirolimus intravenously (IV) on days 1 and 8 or day 1 only and pazopanib hydrochloride orally (PO) daily on days 1-21. Cycles repeat every 21 days until unequivocal clinical disease progression, unacceptable toxicity, or until in the opinion of the investigator the patient is no longer benefiting from therapy, or at the patient's discretion.

After completion of study treatment, participants are followed up at 30 days, then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, >= 18 years old, must have a histologically confirmed diagnosis of non-adipocytic soft tissue sarcoma (STS) that is either metastatic or locally advanced and for which curative therapy is not available, surgery is not a recommended option, and pazopanib treatment is indicated.
* Subjects must have one or more measurable target lesions by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1, assessed via computed tomography (CT) scan or magnetic resonance imaging (MRI).
* Clinical or radiological progression or failure due to toxicity on at least 1 prior regimen of systemic treatment for advanced disease. Subjects may not have received more than 4 prior lines of systemic therapy (no more than 2 prior therapies may be combination cytotoxic therapies). Neo-adjuvant/adjuvant/maintenance treatments are not included for this criterion.
* Last dose of prior therapy must have been completed a minimum of 14 days prior to start of protocol therapy. All ongoing toxicities related to prior therapy must be resolved or grade 1 (except alopecia).

  * NOTE: Toxicities from prior therapy that have resolved with sequelae (e.g. hypothyroidism) and are asymptomatic or well-controlled are not exclusionary.
* Total bilirubin =< upper limit of normal (ULN) mg/dL (Subjects with known Gilbert's syndrome and a total bilirubin =< 3 mg/dl are permitted to enroll to phase 2/expansion phase only with sponsor-investigator approval).
* Aspartate aminotransferase (AST) =< 2.5 x ULN and alanine aminotransferase (ALT) =< 2.5 x ULN.
* Serum creatinine =<1.5 x ULN (If serum creatinine is > 1.5 mg/dL, calculated creatinine clearance > 50 mL/min using the Cockcroft-Gault formula may be included).
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L.
* Platelet count >= 100,000/mm^3 (100 x 10^9/L).
* Hemoglobin >= 9 g/dL.
* Serum triglyceride =< 300 mg/dL.
* Serum cholesterol =< 350 mg/dL.
* Baseline cardiac left ventricular ejection fraction (LVEF) within institutional limits of normal (by echocardiogram or multigated acquisition [MUGA] study).
* Baseline electrocardiogram with corrected QT (QTc) < 480 millisecond (Bazett's).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Male or non-pregnant and non-breast feeding female:

  * Females of child-bearing potential must agree to use highly effective contraception without interruption from initiation of therapy and while on study medication and have a negative serum pregnancy test (beta human chorionic gonadotropin [beta-hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and at the end of study treatment. A highly effective method of contraception is defined as one that results in a low failure rate (that is, < 1% per year), when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner.
  * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study.
* Life expectancy of > 3 months, as determined by the investigator.
* Ability to understand and sign informed consent.
* Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

* Soft tissue sarcomas with biology or defined treatments for which pazopanib is not indicated, including adipocytic STS, gastrointestinal stromal tumors (GIST), or Kaposi's sarcoma.
* Previously received an mTOR (mammalian target of rapamycin) inhibitor or angiogenesis inhibitor.
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases. A subject with controlled and asymptomatic CNS metastases may participate in this study. As such, the patient must have completed any prior treatment for CNS metastases >= 28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
* Subjects with hemoptysis, central nervous system hemorrhage or gastrointestinal hemorrhage within the last 6 months prior to treatment are excluded due to pazopanib-associated risk of bleeding.
* Subjects with severe hepatic impairment and active gastrointestinal bleeding.
* Uncontrolled serious medical or psychiatric illness.
* Subjects with a currently active second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, or other adequately treated carcinoma-in-situ are ineligible. Subjects are not considered to have a currently active malignancy if they have completed therapy and are free of disease for >= 1 year).
* Recent infection requiring systemic anti-infective treatment that was completed =< 14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
* No clinically significant gastrointestinal abnormalities including malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Uncontrolled diabetes mellitus as defined by hemoglobin A1C (HbA1c) > 8% despite adequate therapy.
* Subjects with unstable coronary artery disease, myocardial infarction, or an arterial thromboembolic event during preceding 6 months.
* Subjects with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
* Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of nab-sirolimus. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfenadine) within the 14 days prior to receiving the first dose of nab-sirolimus.
* Active hepatitis B or hepatitis C infection.
* Systemic immunosuppression, including human immunodeficiency virus (HIV) positive status with or without acquired immunodeficiency syndrome (AIDS).
* Subjects with history of intestinal perforations, fistula, hemorrhages and/or hemoptysis =< 6 months prior to first study treatment.
* Subjects with hypercholesterolemia receiving ongoing treatment with simvastatin.
* Subjects who have had major surgery within 28 days of planned initiation of protocol therapy, or patients who have/have had wound dehiscence, or other open wounds (including diabetic or infectious wounds) with active wound complications.
* Subjects with prior history of severe hypersensitivity (grade 3 or higher) to any known drug excipients, including anaphylaxis to human serum albumin.
* Subjects with uncontrolled hypertension, defined as an average systolic blood pressure (SBP) >= 140 mmHg or an average diastolic blood pressure (DBP) >= 90 mmHg despite best supportive care measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Phase II of the study.
Groups:
- Cohort 1, Dose Level 0: Participants received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 4, Dose Level -1: Participants received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 5, Dose Level -2: Participants received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 6, Dose Level 0B: Participants received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 9, Dose Level -1B: Participants received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 10, Dose Level -2B: Participants received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 11, Dose Level 0C: Participants received 30 mg/m^2 of ABI-009 given intravenously on Day 1 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 12, Dose Level 1C: Participants received 45 mg/m^2 of ABI-009 given intravenously on Day 1 of a 21 day cycle, plus daily oral 400 mg of pazopanib
Period: Overall Study
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C
Started | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Completed | 2 | 2 | 2 | 0 | 2 | 1 | 3 | 3
Not Completed | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 19
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30-39 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  40-49 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  50-59 | 1 | 2 | 0 | 0 | 2 | 0 | 2 | 2 | 9
  60-69 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 5
  70 and over | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 11
  Male | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Maximum-tolerated Dose (MTD) of Nab-rapamycin in Combination With Pazopanib (Phase I) - Nab-Rapamycin Dose
Description: Will be estimated using dose-limiting toxicities (DLTs). Will use a Simon's minimax design.
Time Frame: First 2 cycles (3-week cycles, 21 days each)
Population: MTD was determined to be ABI-009 on DAY 1 of a 21 day cycle ONLY in combination with daily oral pazopanib.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received at least one dose of ABI-009: either at 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8, 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8, 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8, 30 mg/m^2 ABI-009 given intravenously on Day 1 only, or 45 mg/m^2 of ABI-009 given intravenously on Day 1 only.
Arm/Group | All Participants
Number analyzed (Participants) | 19
mg/m^2 | 30

2. Primary Outcome: The Maximum-tolerated Dose (MTD) of Nab-rapamycin in Combination With Pazopanib (Phase I) - Pazopanib Dose
Description: Will be estimated using dose-limiting toxicities (DLTs). Will use a Simon's minimax design.
Time Frame: First 2 cycles (3-week cycles, 21 days each)
Population: MTD was determined to be ABI-009 on DAY 1 of a 21 day cycle ONLY in combination with daily oral pazopanib.
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least one dose pazopanib: either daily oral 800 mg of pazopanib, or daily oral 400 mg of pazopanib.
Arm/Group | All Participants
Number analyzed (Participants) | 19
mg | 400

3. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as any Grade 3 or greater adverse event (AE), at least possibly related to either or both nab-sirolimus and pazopanib. Only toxicities with a clearly identified and documented alternative explanation may be deemed non-DLT. Dose-limiting toxicities include any death not clearly due to underlying disease or extraneous causes, or persistent intolerable nonhematologic AE of any grade that requires dose reduction or permanent discontinuation of the study drug, in the opinion of the investigator.
Time Frame: First 2 cycles (3-week cycles, 21 days each)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Dose Level 0: Subjects received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 4, Dose Level -1: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 5, Dose Level -2: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 800 mg of pazopanib
- Cohort 6, Dose Level 0B: Subjects received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 9, Dose Level -1B: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 10, Dose Level -2B: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 11, Dose Level 0C: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 of a 21 day cycle, plus daily oral 400 mg of pazopanib
- Cohort 12, Dose Level 1C: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 of a 21 day cycle, plus daily oral 400 mg of pazopanib
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
Participants | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 2

4. Primary Outcome: Dose Limiting Toxicities
Description: A Dose-limiting toxicity is defined as any Grade 3 or greater adverse event (AE), at least possibly related to either or both nab-Sirolimus or pazopanib. Only toxicities with clearly identified and documented alternative explanation may be deemed non-DLT. Dose-limiting toxicities include any death not clearly due to underlying disease or extraneous causes, or persistent intolerable nonhematologic Ae of any grade that requires dose reduction or permanent discontinuation of the study drug, in the opinion of the investigator.
Time Frame: First 2 cycles (3 week cycles, 21 days each)
Measure: Number; unit: participants
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
participants
  Thrombocytopenia | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2
  Neutropenia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC decreased, Neutropenia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase elevated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Proteinuria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Thrombocytopenia, Oral mucositis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Thrombocytopenia, Neutropenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  No DLT experienced | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1

5. Primary Outcome: Progression-free Survival (PFS) Rate
Description: Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 where progression is defined as a 20% increase in the sum of the longest diameter of target lesions where the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of new lesions. Will be assessed via descriptive statistics.
Time Frame: At 3 months
Population: Three Phase I patients were treated at the recommended Phase II dose of 30 mg/m^2 nab-sirolimus intravenously on Day 1 of a 21-day cycle, with 400 mg of oral daily pazopanib. These three patients were not enrolled in Phase II.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Treatment (ABI-009, Pazopanib): Cohort 11, Dose Level 0C: Participants received 30 mg/m^2 nab-sirolimus intravenously (IV) on Day 1 only and 400 mg of pazopanib hydrochloride orally (PO) daily on days 1-21. Cycles repeat every 21 days until unequivocal clinical disease progression, unacceptable toxicity, or until in the opinion of the investigator the patient is no longer benefiting from therapy, or at the patient's discretion.
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
proportion of participants | 0.33 [0.00 to 0.91]

6. Secondary Outcome: Incidence of Adverse Events Profile
Description: Treatment-related adverse events (AEs) experienced by participants evaluated by Common Terminology Criteria for Adverse Events (CTCAE) 5.0 and determined to be possibly related, probably related, or definitely related to either nab-sirolimus therapy, pazopanib therapy, or both.
Time Frame: Up to 30 days after last dose (an average of 41 weeks)
Measure: Number; unit: adverse events experienced
Groups:
- Cohort 1, Dose Level 0: Subjects received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 800 mg of pazopanib.
- Cohort 4, Dose Level -1: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 800 mg of pazopanib.
- Cohort 5, Dose Level -2: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 800 mg of pazopanib
- Cohort 6, Dose Level 0B: Subjects received 60 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 400 mg of pazopanib.
- Cohort 9, Dose Level -1B: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 400 mg of pazopanib.
- Cohort 10, Dose Level -2B: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 and Day 8 of a 21-day cycle, plus daily oral 400 mg of pazopanib.
- Cohort 11, Dose Level 0C: Subjects received 30 mg/m^2 of ABI-009 given intravenously on Day 1 only of a 21-day cycle, plus daily oral 400 mg of pazopanib.
- Cohort 12, Dose Level 1C: Subjects received 45 mg/m^2 of ABI-009 given intravenously on Day 1 only of a 21-day cycle, plus daily oral 400 mg of pazopanib.
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3
adverse events experienced
  Grade 1 | 34 | 25 | 11 | 16 | 21 | 29 | 15 | 22
  Grade 2 | 30 | 22 | 6 | 16 | 22 | 34 | 8 | 15
  Grade 3 | 10 | 1 | 3 | 8 | 5 | 10 | 0 | 5
  Grade 4 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Median PFS
Description: Will be assessed using RECIST v1.1. Will be assessed via descriptive statistics.
Time Frame: At 6 months
Population: Three Phase I patients were treated at the recommended Phase II dose of 30 mg/m^2 nab-sirolimus intravenously on Day 1 of a 21-day cycle with 400 mg of oral daily pazopanib. These three patients were not enrolled in Phase II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
months | 1.2 [0.79 to NA] — The upper bound of the confidence interval is undefined/infinite due to insufficient number of participants with events.

8. Secondary Outcome: Progression-Free Survival Rate
Description: Will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Will be assessed via descriptive statistics.
Time Frame: At 6 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
proportion of participants | 0.33 [0.00 to 0.91]

9. Secondary Outcome: Median Overall Survival (OS)
Description: Will be summarized using descriptive statistics.
Time Frame: At 12 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
months | 11.1 [5.0 to NA] — The upper bound of the confidence interval is undefined/infinite.

10. Secondary Outcome: Overall Survival
Description: Will be assessed using descriptive statistics.
Time Frame: 12 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
proportion of participants | .33 [0.00 to 0.91]

11. Secondary Outcome: Objective Response Rate (CR + PR)
Description: Will be based on RECIST v1.1. Will be evaluated by CT imaging.
Time Frame: Up to 2 years
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
proportion of participants | 0.00 [0.00 to 0.71]

12. Secondary Outcome: Disease Control Rate (Complete Response [CR] + Partial Response [PR] + Stable Disease [SD])
Description: Will be based on RECIST v1.1evaluated by computed tomography (CT) imaging. Per RECIST V1.1, Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >= 30% decrease in the sum of diameters of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Time Frame: at 24 weeks
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
proportion of participants | 0.33 [0.00 to 0.91]

13. Secondary Outcome: Duration of Response
Description: Will be evaluated by CT imaging.
Time Frame: Up to 2 years
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (ABI-009, Pazopanib)
Number analyzed (Participants) | 3
months | NA [NA to NA] — Since participants did not have a response, we cannot provide duration of response.

ADVERSE EVENTS:
Time Frame: Adverse events are collected continuously from time of consent to 30 days after last dose of study drug (an average of 41 weeks). Duration over which deaths were monitored was from time of consent through study completion, an average of 91 weeks or 21 months.
Description: Systematic assessment of adverse events is completed by regular investigator assessment.
Arm/Group | Cohort 1, Dose Level 0 | Cohort 4, Dose Level -1 | Cohort 5, Dose Level -2 | Cohort 6, Dose Level 0B | Cohort 9, Dose Level -1B | Cohort 10, Dose Level -2B | Cohort 11, Dose Level 0C | Cohort 12, Dose Level 1C
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 1/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/2 | 0/2 | 1/2 | 0/2 | 1/3 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 2/2 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Dose Level 0 (N=2) | Cohort 4, Dose Level -1 (N=2) | Cohort 5, Dose Level -2 (N=2) | Cohort 6, Dose Level 0B (N=2) | Cohort 9, Dose Level -1B (N=2) | Cohort 10, Dose Level -2B (N=3) | Cohort 11, Dose Level 0C (N=3) | Cohort 12, Dose Level 1C (N=3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac disorders, other: Tricuspid valve mass (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Dose Level 0 (N=2) | Cohort 4, Dose Level -1 (N=2) | Cohort 5, Dose Level -2 (N=2) | Cohort 6, Dose Level 0B (N=2) | Cohort 9, Dose Level -1B (N=2) | Cohort 10, Dose Level -2B (N=3) | Cohort 11, Dose Level 0C (N=3) | Cohort 12, Dose Level 1C (N=3)
Platelet Count Decreased (Investigations) | 2 (16) | 1 (3) | 2 (2) | 2 (10) | 2 (4) | 3 (18) | 0 (0) | 2 (11)
Neutrophil Count Decreased (Investigations) | 1 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 1 (1) | 2 (9)
Anemia (Blood and lymphatic system disorders) | 1 (6) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (13) | 1 (1) | 2 (2)
White Blood Cell Decreased (Investigations) | 2 (5) | 2 (3) | 0 (0) | 1 (5) | 2 (4) | 2 (3) | 1 (1) | 2 (3)
Mucositis Oral (Gastrointestinal disorders) | 2 (5) | 2 (3) | 1 (1) | 1 (1) | 1 (6) | 2 (3) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 3 (5)
Fatigue (General disorders) | 2 (5) | 2 (3) | 2 (2) | 1 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 2 (2) | 1 (1) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 2 (3) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Weight Loss (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increase (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection Fraction Decreased (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (7) | 1 (1) | 1 (1) | 0 (0)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flashing Lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations, Other: Platelet Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu Like Symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Hemorrage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Wall PAin (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - other: Palpable bump above Right elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - other: Shoulder and neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis Infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations, other (presumptive viral gastroenteritis - anorexia, nausea, body aches (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinurea (Renal and urinary disorders) | 1 (3) | 0 (0) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic Obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - other: Scalp dermatitis." (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - other: peeling of labial skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
While the study was originally designed as a phase I/II study, only the phase I component of the study was completed..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03660930/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT03660930/ICF_000.pdf